CLINICAL TRIAL: NCT01611909
Title: A Randomised, Double-blinded, Pilot Study Investigating the Safety and Efficacy of Topical P-menthane-3,8-diol Oil Extract in the Treatment of Childhood Impetigo.
Brief Title: Citriodiol® and Impetigo
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Shreya Dixit, Dermatology Research Fellow, Royal North Shore Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Citriodiol®&Impetigo-001
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Impetigo
Keywords: p-menthane-3,8-diol oil extract; topical therapy
MeSH Terms: conditions — Impetigo | interventions — terpin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2% PMDO (Experimental)
  Interventions: Drug: p-menthane-3,8-diol oil
- 5% PMDO (Experimental)
  Interventions: Drug: p-menthane-3,8-diol oil
- Mupirocin (Active Comparator)
  Interventions: Drug: p-menthane-3,8-diol oil

INTERVENTIONS:
Drug: p-menthane-3,8-diol oil — Apply topically to affected area twice daily

SUMMARY:
This study aims to investigate the efficacy and safety of topical p-menthane-3,8-diol (PMD)-rich Corymbia Citriodora oil (Citriodiol®) in children with impetigo. Citriodiol® is already known to be effective as an insect repellent and is safe in its topical application. The investigators have also found in our laboratory that it is bactericidal against Staphylococcus aureus, the bacteria responsible for causing impetigo. Parents are always searching for a natural alternative to antibiotics (the current gold standard treatment for impetigo), and the investigators believe Citriodiol® could provide this possible alternative.

DETAILED DESCRIPTION:
The extract of lemon eucalyptus, a common plant, has since the 1970s been used in commercial insect repellent products. Recently, it has been shown that lemon eucalyptus has potent anti-bacterial and anti-fungal effects that should assist in the treatment of inflammatory conditions such as impetigo. Our aim is to investigate this further by investigating the safety and efficacy of this product in the treatment of Impetigo.

A randomised, double-blinded, three-armed pilot study, involving a total of 30 patients will be recruited from the dermatology outpatient department clinic at Royal North Shore hospital for this study. These patients will be between the ages of 12 months and 12 years with a clinical diagnosis of Impetigo.

The three treatment groups will include a 2% or 5% topical p-menthane-3,8-diol (extracted from lemon eucalyptus) and a topical Mupirocin arm, which will be applied topically twice a day till resolution of symptoms. Follow-up will occur weekly until resolution of symptoms, which is expected within 2 weeks. Photographs, disease severity assessment and lesional swabs for culture will be taken at recruitment and as progress.

ELIGIBILITY:
Inclusion Criteria:

* age between 12 months and 12 years
* dermatologist-confirmed impetigo
* written informed consent provided by parents

Exclusion Criteria:

* impetigo requiring oral/systemic therapy
* diagnosis of another form of staphylococcal or streptococcal disease (eg, cellulitis, erysipelas, abscess)
* serious local infection (eg, cellulitis, abscess, wound infection) or systemic infection
* oral or topical antibiotics
* known allergy to topical insect repellents
* patients receiving systemic corticosteroids, immunosuppressive agents, radiation therapy, chemotherapy within 1 month prior to entry into study
* history of any clinically significant or poorly controlled cardiac, haematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, psychiatric, and/or other major disease as determined by the investigator
* current enrollment in any other trial of an investigational drug within 30 days prior to study drug administration
* other unspecified reasons, in the opinion of the investigator that makes the patient unsuitable for enrollment.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in severity score of impetigo | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia